CLINICAL TRIAL: NCT02000388
Title: Efficacy and Safety of Intranasal Ketorolac Tromethamine (SPRIX) as a Short Term Pain Management Tool for Adult Male Patients With Post-Vasectomy Pain
Brief Title: Intranasal Ketorolac Tromethamine (SPRIX) as a Short Term Pain Management of Post-Vasectomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Citrus Valley Medical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1012-2011-SPRIX
Record Dates: First submitted 2013-11-19; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Post Vasectomy Pain
MeSH Terms: interventions — Ketorolac Tromethamine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac tromethamine (SPRIX) (Other): A SPRIX dose will be one 15.75 mg spray in each nostril for a total dose of 31.5 mg which can be repeated every 6-8 hrs as needed for post vasectomy pain with a maximum daily dose of 126 mg to be continued for up to 5 days.
  Interventions: Drug: Ketorolac Tromethamine
- Standard of care (Other): The intervention used will be standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Ketorolac Tromethamine
  Other Names: SPRIX
  Arms: Ketorolac tromethamine (SPRIX)
Other: Standard of Care
  Arms: Standard of care

SUMMARY:
To evaluate the efficacy, tolerability and safety of intranasal ketorolac tromethamine (SPRIX) as an option for pain management in post vasectomy patients.

ELIGIBILITY:
INCLUSION CRITERIA

1. Male Subject must be between the age twenty five (25) years and sixty four (64)
2. Willing and able to provide an informed consent
3. Has made decision to undergo vasectomy
4. Subject is in good general physical condition as assessed by the Principal Investigator

EXCLUSION CRITERIA

1. Current treatment with or known allergy or sensitivity to all forms of ketorolac tromethamine , aspirin , other non steroidal anti inflammatory drugs (NSAIDs) or Ethylenediaminetetraacetic acid (EDTA)
2. Use of narcotics/opiate or medical marijuana within one (1) week prior to the baseline visit and entire study participation
3. Use of illegal drugs by self reporting
4. History of drug or alcohol abuse within five (5) years of screening visit
5. History of suicide attempt within five (5) years of screening visit
6. A diagnosis of a severe neuro-psychiatric disease
7. Subject who is currently receiving investigational drug(s) or participated in a clinical trial involving investigational drug(s) within thirty (30) day of the screening visit
8. Subject with history of any of the following coronary conditions: (chronic stable angina being currently treated with long acting nitrates, chronic stable angina require treatment with short acting nitrates with 90 days of visit 1, angina occurring during sexual intercourse in the last six months, unstable angina within six months of visit 1
9. Resting, sitting blood pressure (BP) > 160mm Hg in systolic pressure or > 100mm Hg is diastolic pressure at screening. If a patient is found to have untreated significant hypertension at screening and antihypertensive treatment is initiated, assessment for study eligibility should be deferred until BP and antihypertensive medication have been stable for at least one month. For patients with previously diagnosed hypertension, antihypertensive medications must be stable for at least one month prior to screening.
10. Known or suspected cerebrovascular bleeding, hemorrhagic diathesis or incomplete hemostasis, and those at high risk of bleeding, have history of a bleeding problem or low platelet count or coagulation disorder or are on therapy that affects homeostasis
11. Active peptic ulcer disease, recent GI bleeding or perforation, or a history of peptic ulcers or GI bleeding
12. History of asthma, urticaria or other allergic-type reaction after taking aspirin or other non steroidal inflammatory drugs (NASIDs)
13. Subject over sixty four (64) years of age
14. Subject with any clinically significant renal function or liver abnormality
15. Subject who has history of swelling of face, mouth, tongue, lips, gums, neck, or throat (angioedema) or with cardiac decompensation or similar conditions
16. Major surgery scheduled within 3 weeks or screening and for entire participation of study
17. Current exfoliative dermatitis, Stevens-Johnson syndrome or toxic epidermal necrolysis
18. Any condition in the opinion of the investigator that makes the subject unsuitable for study

    -

Ages: 25 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 5 days

SECONDARY OUTCOMES:
To determine Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Edward L Davis, M.D., Principal Investigator — Citrus Valley Medical Research, Inc.